CLINICAL TRIAL: NCT00412737
Title: A Double-blind, Randomized, Placebo Controlled, Multi-center Trial of Oseltamivir for the Seasonal Prophylaxis of Influenza in Immunocompromised Patients
Brief Title: A Study of Oseltamivir (Tamiflu) for the Seasonal Prophylaxis of Influenza in Immunocompromised Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NV20235
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Results first posted 2009-09-09 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oseltamivir (Experimental)
  Interventions: Drug: Oseltamivir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir 30 mg to 75 mg capsule or suspension orally once daily for 12 weeks.
  Other Names: Tamiflu
  Arms: Oseltamivir
Drug: Placebo — Placebo matched to oseltamivir capsule or suspension orally once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
This 2 arm study will evaluate the efficacy and safety of oseltamivir in the seasonal prophylaxis of influenza in immunocompromised participants (as represented by transplant recipients). Transplant recipients enrolled when influenza is circulating in the community will be randomized to receive oseltamivir syrup or capsules 30 milligrams (mg) to 75 mg daily (depending on body weight) or placebo for 12 weeks. Influenza symptoms and safety data will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Negative rapid diagnostic test for influenza at baseline;
* Immunocompromised participant (liver and/or kidney recipient or allogenic hematopoietic stem cell transplant).

Exclusion Criteria:

* Symptoms suggestive of influenza-like illness; but not limited to fever, cough, or nasal congestion;
* Influenza vaccination in 6 weeks prior to randomization;
* Positive rapid diagnostic test for influenza;
* Solid organ transplant within 6 months of randomization;
* Antiviral treatment for influenza in 2 weeks prior to randomization.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (69):
- United States (31):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Stanford, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Newark, Delaware
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Brooklyn Center, Minnesota
  - Missoula, Montana
  - Camden, New Jersey
  - Hackensack, New Jersey
  - Livingston, New Jersey
  - Newark, New Jersey
  - Buffalo, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
- Belgium (4):
  - Aalst
  - Brussels
  - Edegem
  - Leuven
- Canada (5):
  - Edmonton, Alberta
  - Coquitlam, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Saskatoon, Saskatchewan
- Brno, Czechia
- Estonia (2):
  - Tallinn
  - Tartu
- France (3):
  - Paris
  - Toulouse
  - Tours
- Germany (5):
  - Aachen
  - Berlin
  - Hamburg
  - Heidelberg
  - München
- Hungary (3):
  - Budapest
  - Pécs
  - Szeged
- Israel (3):
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Italy (3):
  - Padua
  - Pavia
  - Roma
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (4):
  - Bialystok
  - Lodz
  - Szczecin
  - Warsaw
- Madrid, Spain
- United Kingdom (2):
  - Birmingham
  - Edinburgh

REFERENCES:
- [Derived] Ison MG, Szakaly P, Shapira MY, Krivan G, Nist A, Dutkowski R. Efficacy and safety of oral oseltamivir for influenza prophylaxis in transplant recipients. Antivir Ther. 2012;17(6):955-64. doi: 10.3851/IMP2192. Epub 2012 Jun 22. PMID 22728756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of total 477 participants who were randomized to receive study treatments, 2 participants were not included in the study population due to lack of efficacy data. Thus, results are reported only for 475 participants.
Pre-assignment Details: One participant was randomized to placebo group but received oseltamivir for the first 9 weeks of the study. This participant was included in the placebo group in the Intention-to-treat (ITT) analysis population, but in the oseltamivir group in the safety analysis population.
Groups:
- Oseltamivir: Oseltamivir 30 milligram (mg) to 75 mg capsule or suspension orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Oseltamivir
Started | 237 | 238
Completed | 221 | 232
Not Completed | 16 | 6
Not completed — Death | 1 | 0
Not completed — Adverse Event | 3 | 2
Not completed — Refused Treatment | 6 | 2
Not completed — Failure to Return | 6 | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug and had at least 1 post baseline safety assessment. Participants were analyzed as per actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Oseltamivir | Total
Number analyzed (Participants) | 237 | 238 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (15.67) | 49.4 (15.47) | 49.2 (15.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 74 | 160
  Male | 151 | 164 | 315

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Laboratory-Confirmed Clinical Influenza, ITT Population
Description: Laboratory-confirmed clinical influenza was defined as a fever (oral or otic temperature greater than [>] 37.2 degrees Celsius [°C]) and a symptom score for cough and/or coryza (nasal congestion on the diary cards, where 0=absent, 1=mild, 2=moderate, and 3=severe) of 1, 2 or 3 on the same day as fever, and laboratory confirmation of influenza either by detection of viral shedding by viral culture from nasopharyngeal swabs within two days of fever and symptoms, and/or by 4-fold or greater increase in serum hemagglutination inhibition (HAI) titers measured from baseline to any point during the study.
Time Frame: From baseline up to 28 days after the last dose of study drug (maximum up to 112 days)
Population: ITT population included all randomized participants who received at least 1 dose of study drug and had at least 1 post baseline efficacy assessment. Participants were analyzed as per initial randomization.
Measure: Number; unit: participants
Arm/Group | Placebo | Oseltamivir
Number analyzed (Participants) | 238 | 237
participants | 7 | 5
Statistical Analysis 1: Comparison: Placebo vs Oseltamivir; The null hypothesis tested was that there was no difference between the proportions of participants who met the primary endpoint in the two treatment groups; Test type: Superiority or Other; p = 0.772, Fisher Exact; Relative Risk Reduction = 0.283, 95% CI 2-sided [-2.3 to 4.1] — Relative Risk Reduction = (1.0 - Relative Risk)

2. Secondary Outcome: Number of Participants With Laboratory Confirmed Clinical Influenza, Per Protocol (PP) Population
Description: Laboratory-confirmed clinical influenza was defined as a fever (oral or otic temperature greater than 37.2 °C) and a symptom score for cough and/or coryza (nasal congestion on the diary cards, where 0=absent, 1=mild, 2=moderate, and 3=severe) of 1, 2 or 3 on the same day as fever, and laboratory confirmation of influenza either by detection of viral shedding by viral culture from nasopharyngeal swabs within two days of fever and symptoms, and/or by 4-fold or greater increase in serum HAI titers measured from baseline to any point during the study.
Time Frame: From baseline up to 28 days after the last dose of study drug (maximum up to 112 days)
Population: Per-Protocol (PP) population was defined as the subset of the ITT population who did not have any major protocol violations which would impact the assessment of efficacy.
Measure: Number; unit: participants
Arm/Group | Placebo | Oseltamivir
Number analyzed (Participants) | 208 | 220
participants | 6 | 4
Statistical Analysis 1: Comparison: Placebo vs Oseltamivir; Test type: Superiority or Other; p = 0.534, Fisher Exact; Relative Risk Reduction = 0.37, 95% CI 2-sided [-2.1 to 4.5] — Relative Risk Reduction = (1.0 - Relative Risk)

3. Secondary Outcome: Number of Participants With Laboratory Confirmed Clinical Influenza, Intent-to-treat Virus Negative at Baseline (ITTNAB) Population
Description: as for outcome 2
Time Frame: From baseline up to 28 days after the last dose of study drug (maximum up to 112 days)
Population: ITTNAB population was defined as the subset of the ITT population who were culture negative at baseline.
Measure: Number; unit: participants
Arm/Group | Placebo | Oseltamivir
Number analyzed (Participants) | 231 | 232
participants | 7 | 4
Statistical Analysis 1: Comparison: Placebo vs Oseltamivir; Test type: Superiority or Other; p = 0.381, Fisher Exact; Relative Risk Reduction = 0.431, 95% CI 2-sided [-1.7 to 4.6] — Relative Risk Reduction = (1.0 - Relative Risk)

4. Secondary Outcome: Number of Participants With Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) Confirmed Clinical Influenza, ITT Population
Description: RT-PCR confirmed clinical influenza was defined as a confirmation of influenza by positive RT-PCR result within 2 days of symptoms/last dose from baseline to any point during the study.
Time Frame: From baseline up to 28 days after the last dose of study drug (maximum up to 112 days)
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Placebo | Oseltamivir
Number analyzed (Participants) | 238 | 237
participants | 7 | 2
Statistical Analysis 1: Comparison: Placebo vs Oseltamivir; Test type: Superiority or Other; Relative Risk Reduction = 0.713, 95% CI 2-sided [-0.6 to 5.2] — Relative Risk Reduction = (1.0 - Relative Risk)

5. Secondary Outcome: Number of Participants With RT-PCR Confirmed Clinical Influenza, ITTNAB Population
Description: as for outcome 4
Time Frame: From baseline up to 28 days after the last dose of study drug (maximum up to 112 days)
Population: ITTNAB population.
Measure: Number; unit: participants
Arm/Group | Placebo | Oseltamivir
Number analyzed (Participants) | 231 | 232
participants | 7 | 1
Statistical Analysis 1: Comparison: Placebo vs Oseltamivir; Test type: Superiority or Other; Slope = 0.858, 95% CI 2-sided [0.1 to 5.7] — Relative Risk Reduction = (1.0 - Relative Risk)

6. Secondary Outcome: Number of Participants With RT-PCR, or Serology/Viral Culture Confirmed Clinical Influenza, ITT Population
Description: RT-PCR, or serology/viral culture confirmed clinical influenza was defined as a confirmation of influenza by positive RT-PCR or culture within 2 days of symptoms/ last dose and/or positive serology result from baseline to any point during the study.
Time Frame: From baseline up to 28 days after the last dose of study drug (maximum up to 112 days)
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Placebo | Oseltamivir
Number analyzed (Participants) | 238 | 237
participants | 8 | 5
Statistical Analysis 1: Comparison: Placebo vs Oseltamivir; Test type: Superiority or Other; Relative Risk Reduction = 0.372, 95% CI 2-sided [-1.9 to 4.6] — Relative Risk Reduction = (1.0 - Relative Risk)

7. Secondary Outcome: Number of Participants With RT-PCR, or Serology/Viral Culture Confirmed Clinical Influenza, ITTNAB Population
Description: as for outcome 6
Time Frame: From baseline up to 28 days after the last dose of study drug (maximum up to 112 days)
Population: ITTNAB population.
Measure: Number; unit: participants
Arm/Group | Placebo | Oseltamivir
Number analyzed (Participants) | 231 | 232
participants | 8 | 4
Statistical Analysis 1: Comparison: Placebo vs Oseltamivir; Test type: Superiority or Other; Relative Risk Reduction = 0.502, 95% CI 2-sided [-1.4 to 5.1] — Relative Risk Reduction = (1.0 - Relative Risk)

ADVERSE EVENTS:
Time Frame: From baseline up to 2 days after the last dose of study drug (maximum up to 86 days)
Description: Safety population.
Arm/Group | Placebo | Oseltamivir
Serious Adverse Events (participants affected / at risk) | 23/237 | 18/238
Other Adverse Events (participants affected / at risk) | 40/237 | 42/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=237) | Oseltamivir (N=238)
Gastroenteritis (Infections and infestations) | 1 | 4
Pneumonia (Infections and infestations) | 3 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thalamus haemorrhage (Nervous system disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Nephropathy (Renal and urinary disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug interaction (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Acute graft versus host disease (Immune system disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=237) | Oseltamivir (N=238)
Diarrhoea (Gastrointestinal disorders) | 18 | 15
Headache (Nervous system disorders) | 12 | 11
Nausea (Gastrointestinal disorders) | 9 | 13
Fatigue (General disorders) | 7 | 12

LIMITATIONS AND CAVEATS:
There were no overall limitations and caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.